CLINICAL TRIAL: NCT06794398
Title: Feasibility of Appropriate Smartphone Position During Video-assisted Cardiopulmonary Resuscitation When the Bystander is Alone At the Scene - a Randomized Controlled Crossover Simulation Trial
Brief Title: Feasibility of Appropriate Smartphone Position During Video-assisted Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr. Bálint Bánfai, associate professor, University of Pecs
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: V-CPR alone at the scene
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: video-assisted cardiopulmonary resuscitation; cardiac arrest; cardiopulmonary resuscitation; lay responder
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- V-CPR in the room (Experimental): Participants should perform a simulated V-CPR scenario based on the European Resuscitation Council 2021 Guidelines in a prepared room (inside environment).
  Interventions: Device: V-CPR inside a room when the lay responder is alone (no operator for holding the phone); Device: V-CPR in a yard (outside environment) when the lay responder is alone (no operator for holding the phone)
- V-CPR outside (Experimental): Participants should perform a simulated V-CPR scenario based on the European Resuscitation Council 2021 Guidelines in a prepared yard (outside environment).
  Interventions: Device: V-CPR inside a room when the lay responder is alone (no operator for holding the phone); Device: V-CPR in a yard (outside environment) when the lay responder is alone (no operator for holding the phone)

INTERVENTIONS:
Device: V-CPR inside a room when the lay responder is alone (no operator for holding the phone) — Participants should find an appropriate smartphone position when they were able to use any objects in their environment. Participants get video-based (vocal and visual) instructions from the dispatcher during the V-CPR situation.
Device: V-CPR in a yard (outside environment) when the lay responder is alone (no operator for holding the phone) — Participants should find an appropriate smartphone position when they were able to use any objects in their environment. Participants get video-based (vocal and visual) instructions from the dispatcher during the V-CPR situation.

SUMMARY:
There is a gap in our knowledge regarding whether video-assisted cardiopulmonary resuscitation (V-CPR) is feasible when a lay responder is alone at the scene. The feasibility of V-CPR was measured in a simulated cardiac arrest scenario when a lay responder was alone with the patient.

DETAILED DESCRIPTION:
There is a gap in our knowledge regarding whether video-assisted cardiopulmonary resuscitation (V-CPR) is feasible when a lay responder is alone. The feasibility of V-CPR was measured in a simulated cardiac arrest scenario when a lay responder was alone with the patient. A pilot study was conducted to measure the appropriate smartphone position and placement time when a lay responder is alone. Two simulated cardiac arrest locations were prepared: a living room and yard.

The performance of the participants were recorded. After that, the quality and assessability of the videos were evaluated by five experts (experienced in CPR teaching and evaluation).

ELIGIBILITY:
Inclusion Criteria:

* layperson or health care professional, who is phisically and mentally able to do a simulated CPR scenario (participants in the scenario)
* expert in CPR training (assessors)

Exclusion Criteria:

* technical issue during data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Smartphone camera placement and perspective (used objects and visible environment) | During procedure
  Evaluating the used object (chair, table, shue, etc) to stabilize the smartphone for V-CPR in the prepared environment (a photo was taken by the study operator).
  Evaluating smartphone camera perspective by the dispatcher's laptop screen (smartphone camera picture was transferred via Microsoft Teams from the smartphone to the laptop during a live video-stream (to see what the dispatcher did see). Live video-stream was also recorded for post-analysis.

SECONDARY OUTCOMES:
Smartphone camera placement time (time to the first chest compression) | During procedure
  Measuring the time from the dispatcher's instructions to the first chest compression (putting the hand on the patient's chest) based on the recorded video.

OTHER OUTCOMES:
General quality of the video-records (clarity, lagging, camera perspective, visibility of chest compressions; by using a Likert-scale: from "1 - very bad quality" to "4 - very good quality") | During post-analysis of the video-records (within 1 week after data collection)
  Measuring the general quality of the video-records (Is chest compression depth, rate and hand position visible?; clarity and lagging of the video-record) based on the assessors subjective answers by using a Likert-scale: from "1 - very bad quality" to "4 - very good quality").

CONTACTS AND LOCATIONS:
Overall Officials: Bálint Bánfai, Ph.D, Principal Investigator — University of Pecs
Locations (1):
- Human Patient Simulation Center, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banfai B, Betlehem J, Jobb B, Horvath B, Mate-Pohr K, Nemeth D, Musch J, Banfai-Csonka H. Feasibility of video-assisted cardiopulmonary resuscitation when the lay responder is alone with the victim: a randomized controlled crossover pilot study. Sci Rep. 2025 Jul 19;15(1):26268. doi: 10.1038/s41598-025-12014-6. PMID 40683935